CLINICAL TRIAL: NCT01620190
Title: A Phase II Study of Weekly Abraxane for Patients With Advanced NSCLC With EGFR Mutations or With Durable Response to an EGFR Tyrosine Kinase Inhibitor Following Front Line Therapy With EGFR Tyrosine Kinase Inhibitors
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Previously Treated Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Christina S Baik, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7755; NCI-2012-00865 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7755 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1712044 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (paclitaxel albumin-stabilized nanoparticle formula) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; nab-paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; protein-bound paclitaxel

SUMMARY:
This research study examines the use of Abraxane (paclitaxel albumin-stabilized nanoparticle formulation) in patients with lung cancer. Abraxane is a chemotherapy approved to treat patients with breast cancer. Doctors want to know if Abraxane is safe and effective in treating patients with lung cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) and epidermal growth factor receptor (EGFR) mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate of weekly nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) in patients with advanced non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutations following front-line therapy with EGFR tyrosine kinase inhibitors (TKI).

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of weekly nab-paclitaxel in patients with advanced NSCLC with EGFR mutations following front-line therapy with an EGFR TKI.

II. To evaluate the time-to-progression and overall survival.

OUTLINE:

Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer with documented EGFR mutation in tumor deoxyribonucleic acid (DNA) or complete/partial response to first line EGFR tyrosine kinase inhibitors with > or = to 6 months duration of response in patients who do not have a confirmed EGFR mutation
* At least one site of measurable disease as determined by the Investigator, using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Progressive disease with radiographic evidence of disease progression per investigator assessment during therapy with an EGFR tyrosine kinase inhibitor in the metastatic setting; patients may continue EGFR inhibitor therapy throughout the screening period until the day prior to nab-paclitaxel treatment initiation
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 at the time of informed consent
* Platelet count >= 100,000/uL
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 9 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) = < 2.5 times upper limit of normal
* Alkaline phosphatase =< 2.5 times upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Bilirubin =< 1.5 mg/dL
* Creatinine =< 1.5 mg/dL
* Women of child-bearing potential (WOCP) and sexually active men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, during treatment and for three months after completing treatment
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of childbearing potential
* Life expectancy of > 12 weeks
* Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

* Prior conventional cytotoxic chemotherapy for metastatic or recurrent disease; prior adjuvant, neoadjuvant or chemoradiotherapy for NSCLC is permitted, provided at least 6 months elapsed prior to documented metastatic recurrence
* A single dose of a platinum doublet discontinued due to intolerability without evidence of disease progression is permitted
* Patient is < 5 years free of another primary malignancy, except: a) if the other malignancy is basal cell carcinoma or cervical carcinoma in situ or b) if the other primary malignancy is not considered clinically significant and is requiring no active intervention
* Progressive or symptomatic central nervous system (CNS) metastases; patients with known brain metastasis must have stable disease following treatment with surgery, radiation or both; in addition, they must be off corticosteroids
* Radiotherapy within 7 days of study treatment
* Peripheral neuropathy grade 2 or greater
* Grade III/IV congestive heart failure, as defined by New York Heart Association (NYHA) criteria, or myocardial infarction within 6 months
* Any serious or uncontrolled concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
* Patient has known chronic liver disease, e.g. diagnosis of chronic active hepatitis or cirrhosis
* Major surgery within 21 days of study treatment; minor surgery within 2 weeks of study treatment; placement of vascular access device and biopsies allowed and is not considered major or minor surgery
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Pregnant or breast feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12-02 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2019-04-29

CONTACTS AND LOCATIONS:
Overall Officials: Christina Baik, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (12):
- United States (12):
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Group Health Cooperative, Redmond, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seattle Cancer Care Alliance Network Office/University of Washington Phase II open label study enrolled patients at five sites between December 2012 and April 2017.
Pre-assignment Details: Twenty-six patients were consented and treated.
Period: Overall Study
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participant measures are based on total eligible, consented, and treated patients.
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 65 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Response) Defined by RECIST 1.1 Criteria
Description: The response rate as the proportion and 95% confidence interval of patients who achieved a complete response or partial response will be calculated.
Time Frame: Assessed every two cycles from date of first study therapy until documented disease progression, date of death, unacceptable toxicity, or withdrawal of patient consent, whichever occurs first, assessed up to 60 weeks.
Population: All participants who met eligibility criteria and received at least one dose of study intervention and at least one assessment post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 26
Participants
  Complete Response | 0
  Partial Response | 9
  Stable Disease | 6
  Progressive Disease | 6
  Not Evaluable | 5

2. Secondary Outcome: Overall Percentage of Patients Experiencing Toxicity Within a Clinically Significant Category Defined as Neutropenia, Neutropenic Fever, or Neuropathy.
Description: Toxicity rates will be described as percentage of patient who experienced a Grade 3 or higher clinically significant toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Collected from the time patient received the first dose of study therapy through 30 days following the last dose of study therapy or the start of a new cancer therapy, whichever occurred first, assessed up to 64 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 26
Participants | 4

3. Secondary Outcome: Overall Survival
Description: Will report as median values with their respective 95% confidence intervals will be reported. Time to event distribution will be estimated using Kaplan-Meier method.
Time Frame: Assessed from date of patient consent until date of death from any cause or withdrawal of patient consent, whichever occurs first, assessed up to 305 weeks.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 26
weeks | 36 [16.8 to 68]

4. Secondary Outcome: Overall Percentage of Patients Experiencing Grade 3 or Higher Toxicity.
Description: Toxicity rates will be described as percentage of patients experiencing Grade 3 or higher toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 26
Participants | 8

5. Secondary Outcome: Time to Progression.
Description: Reported as median values with their respective 95% confidence intervals for patients who were assessed. Time to event distribution will be estimated using the Kaplan-Meier method.
Time Frame: Assessed from date of patient consent until documented disease progression, date of death from any cause, start of new anti-cancer therapy, or withdrawal of patient consent, whichever occurs first, assessed up to 60 weeks.
Population: 10 patients were not included in the confidence interval as 5 patients passed away before documented radiological Progressive Disease could be assessed and 5 patients initiated new therapy before documented radiological Progressive Disease could be assessed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
Number analyzed (Participants) | 16
weeks | 10.2 [3.4 to 60.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time patient received the first dose of study therapy through 30 days following the last dose of study therapy or the start of a new cancer therapy, assessed up to to 64 weeks. All-Cause Mortality was assessed up to 305 weeks.
Description: Any adverse events leading to a treatment interruption or dose reduction along with all adverse events that are grade 3 and higher were recorded.
Arm/Group | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula)
All-Cause Mortality (participants affected / at risk) | 6/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula) (N=26)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel Albumin-stabilized Nanoparticle Formula) (N=26)
Fatigue (General disorders) | 4 (4)
Peripheral Neuropathy (Nervous system disorders) | 6 (7)
Neutrophil count decreased (Investigations) | 4 (5)
White blood cell decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT01620190/Prot_SAP_000.pdf